CLINICAL TRIAL: NCT01931787
Title: A Pilot Clinical Trial of CPI-613 in Patients With Relapsed or Refractory Small Cell Lung Carcinoma (SCLC)
Brief Title: CPI-613 in Treating Patients With Relapsed or Refractory Small Cell Lung Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00024405; NCI-2013-01653 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CCCWFU 62113 (Other: Comprehensive Cancer Center of Wake Forest University); P30CA012197 (NIH)
Record Dates: First submitted 2013-08-27; First posted 2013-08-29 (Estimated); Last update posted 2018-07-03 (Actual); Status verified 2018-07

CONDITIONS: Recurrent Small Cell Lung Cancer
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — devimistat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (CPI-613) (Experimental): Patients receive CPI-613 IV over 2 hours on days 1 and 4 of weeks 1-3. Courses repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: 6,8-bis(benzylthio)octanoic acid

INTERVENTIONS:
Drug: 6,8-bis(benzylthio)octanoic acid — Given IV
  Other Names: alpha-lipoic acid analogue CPI-613; CPI-613

SUMMARY:
This pilot clinical trial studies CPI-613 (6,8-bis[benzylthio]octanoic acid) in treating patients with relapsed or refractory small cell lung cancer. CPI-613 may interfere with the growth of tumor cells and may be an effective treatment for small cell lung cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the safety and anti-cancer activities in patients with relapsed or refractory small cell lung cancer (SCLC) who have failed 1 or 2 lines of chemotherapy.

OUTLINE:

Patients receive CPI-613 intravenously (IV) over 2 hours on days 1 and 4 of weeks 1-3. Courses repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 2 months.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically proven SCLC that has relapsed or been refractory from at least one line of chemotherapy
* Eastern Cooperative Oncology Group (ECOG) performance status of =< 3
* Expected survival > 1 month
* No acute toxicities from previous treatment higher than grade 1 at the start of treatment with CPI-613
* Women of child-bearing potential (i.e., women who are pre-menopausal or not surgically sterile) must use accepted contraceptive methods (abstinence, intrauterine device [IUD], oral contraceptive or double barrier device) during the study, and must have a negative serum or urine pregnancy test within 1 week prior to treatment initiation
* Men must practice effective contraceptive methods during the study, unless documentation of infertility exists
* Platelet count >= 100,000 cells/mm^3 or >= 100 bil/L
* Absolute neutrophil count (ANC) >= 1500 cells/mm^3 or >= 1.5 bil/L
* Aspartate aminotransferase (AST/serum glutamic oxaloacetic transaminase [SGOT]) =< 3 x upper normal limit (UNL)
* Bilirubin =< 1.5 x UNL
* Serum creatinine =< 1.5 mg/dL or 133 µmol/L
* Albumin > 2.0 g/dL or > 20 g/L
* Mentally competent, ability to understand and willingness to sign an Institutional Review Board (IRB)-approved written informed consent form
* Have access via central line (e.g., portacath)-double lumen due to CPI-613 administration requirements

Exclusion Criteria:

* Patients receiving any other standard or investigational treatment for their cancer, or any investigational agent for any non-cancer indication within the past 2 weeks prior to initiation of CPI-613 treatment
* Serious medical illness that would potentially increase patients' risk for toxicity
* Any active uncontrolled bleeding or bleeding diathesis
* Pregnant women, women of child-bearing potential not using reliable means of contraception, or lactating women
* Men unwilling to practice contraceptive methods during the study period
* Life expectancy less than 1 month
* Treatment with any anti-cancer therapy within the 2 weeks prior to treatment with CPI-613
* Patients with untreated central nervous system (CNS) or epidural tumor
* Any condition or abnormality which may, in the opinion of the investigator, compromise his or her safety
* Unwilling or unable to follow protocol requirements
* Active heart disease including myocardial infarction within previous 6 months, symptomatic coronary artery disease, arrhythmias not controlled with medication, or symptomatic congestive heart failure
* Evidence of active infection or serious infection (e.g., septic shock with multi-organ dysfunction) within the past month
* Patients with known human immunodeficiency virus (HIV) infection
* Requirement for immediate palliative treatment of any kind including surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2013-10 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Tumor response rates, defined as the proportion of patients who achieve complete response (CR), partial response (PR), stable disease (SD) or progressive disease (PD) | Up to 3 years
  The proportion of responders as the percent of patients who are SD, PR and CR will be estimated, as well as RR (sum of PR + CR) and disease control rate (DCR, which is the sum of SD, PR and CR). 95% confidence intervals will be included.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | Up to 3 years
  Survival curves for PFS will be estimated using Kaplan-Meier techniques. In addition, the 6 month and 1-year PFS rates will be estimated. Median PFS will be estimated as well.
Overall survival (OS) | Up to 3 years
  Survival curves for OS will be estimated using Kaplan-Meier techniques. In addition, the 6 month and 1-year OS rates will be estimated. Median OS will be estimated as well.

OTHER OUTCOMES:
Incidence of toxicities, graded according to the Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 | Up to 3 years
  Each toxicity identified in the protocol will be examined by grade.

CONTACTS AND LOCATIONS:
Overall Officials: Jimmy Ruiz, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Comprehensive Cancer Center of Wake Forest University, Winston-Salem, North Carolina, United States